CLINICAL TRIAL: NCT00003811
Title: High-Dose Cisplatin, Etoposide and Bleomycin (HD-PEB) Combined With Amifostine in Children With High-Risk Malignant Germ Cell Tumors - A POG Pilot Study
Brief Title: Combination Chemotherapy Plus Amifostine in Treating Children With Malignant Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 9749; POG-9749 (Other: Pediatric Oncology Group); CDR0000066956 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-12-10 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Childhood Germ Cell Tumor; Drug/Agent Toxicity by Tissue/Organ; Extragonadal Germ Cell Tumor; Ovarian Cancer
Keywords: drug/agent toxicity by tissue/organ; childhood teratoma; childhood malignant testicular germ cell tumor; childhood malignant ovarian germ cell tumor; childhood extragonadal germ cell tumor; recurrent childhood malignant germ cell tumor
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Ovarian Neoplasms; Teratoma; Testicular Neoplasms; Ovarian Germ Cell Cancer | interventions — Bleomycin; Amifostine; Cisplatin; Etoposide

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: amifostine trihydrate
Drug: cisplatin
Drug: etoposide
Procedure: conventional surgery

SUMMARY:
RATIONALE: Chemotherapy drugs use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs such as amifostine may protect normal cells from the side effects of chemotherapy.

PURPOSE: Phase I trial to study the effectiveness of high-dose cisplatin, etoposide, and bleomycin plus amifostine in treating children who have malignant germ cell tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the early efficacy and toxicity profile of high-dose cisplatin, etoposide, bleomycin, and amifostine in children with newly diagnosed, high-risk malignant, extragonadal germ cell tumors. II. Determine whether the use of amifostine can reduce the hematologic and nonhematologic toxic effects of this combination chemotherapy in these patients when compared to similar patients treated on POG-9049/CCG-8881 with the same combination chemotherapy. III. Determine the response rate of patients treated with this regimen.

OUTLINE: Patients undergo surgical biopsy or resection. Patients then receive bleomycin IV over 10 minutes on day 1 and etoposide IV over 1 hour, amifostine IV over 15 minutes, and cisplatin IV over 1 hour on days 1-5. Treatment repeats every 3-4 weeks for 4 courses in the absence of unacceptable toxicity or disease progression. Patients who have no disease after 4 courses of chemotherapy receive no further treatment. Patients who have residual disease undergo second-look surgery. After surgery, patients who still have active tumor receive 2 additional courses of chemotherapy. Those patients who still have tumor after the 2 additional courses may have a third surgery. Patients are followed every month for 6 months, every 2 months for 6 months, every 6 months for 1 year, and then annually thereafter until death.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study within 1.39 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed, newly diagnosed, high-risk, extracranial germ cell tumors including the following: Yolk sac carcinoma (endodermal sinus tumor) Embryonal carcinoma Choriocarcinoma Teratoma with mixed malignant elements (malignant teratoma) OR Malignant recurrence (stage III or IV) of previously resected stage I extracranial, extragonadal tumor High-risk disease defined as stage III or IV extragonadal tumors Measurable disease by diagnostic imaging

PATIENT CHARACTERISTICS: Age: Under 15 at time of diagnosis Performance status: Not specified Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 750/mm3 Platelet count greater than 75,000/mm3 Hepatic: Not specified Renal: Creatinine normal OR Glomerular filtration rate at least 50% of normal

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2000-04; Primary Completion 2004-10 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Feasibility from Efficacy Standpoint
  The hazard rate is constant over 1.39 years, then the probability of the occurrence of a failure within this time interval follows a Poisson distribution. The table below shows the trial feasibility probabilities associated with those failure rates. We define the probability of feasibility as the probability of observing a total of at most less than three failures in 25 patient years of follow-up.

SECONDARY OUTCOMES:
Assessment of Reduction in Toxicity
  Descriptive statistics will be performed for nephrotoxicity, hematologic and pulmonary toxicities, and inference will be performed for ototoxicity. Frequency tables of the occurrences of toxicities by grade will be tabulated for ANC and platelets. To assess nephrotoxicity and pulmonary toxicity, descriptive statistics will be calculated for GFR and DLCO, respectively. These statistics will be compared to the corresponding summaries on the appropriate population of patients from POG 9049/CCG 8881.

CONTACTS AND LOCATIONS:
Overall Officials: Neyssa M. Marina, MD, Study Chair — Stanford University
Locations (110):
- United States (97):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - Children's Hospital and Health Center, San Diego, California
  - Naval Medical Center - San Diego, San Diego, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Stanford University Medical Center, Stanford, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Walt Disney Memorial Cancer Institute, Orlando, Florida
  - CCOP - Florida Pediatric, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Hope Children's Hospital, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Portland, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - St. John's Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - University of Missouri-Columbia Hospital and Clinics, Columbia, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Mission Saint Joseph's Health System, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Oklahoma Memorial Hospital, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - James H. Quillen College of Medicine, Johnson City, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - MBCCOP - South Texas Pediatric, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Clinic, Temple, Texas
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Carilion Roanoke Community Hospital, Roanoke, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Medical School-Charleston, Charleston, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Royal Children's Hospital, Parkville, Victoria, Australia
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier de L'Universite Laval, Sainte-Foy, Quebec
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- San Jorge Childrens Hospital, Santurce, Puerto Rico
- Switzerland (2):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Clinique de Pediatrie, Geneva

REFERENCES:
- [Result] Marina N, Chang KW, Malogolowkin M, London WB, Frazier AL, Womer RB, Rescorla F, Billmire DF, Davis MM, Perlman EJ, Giller R, Lauer SJ, Olson TA; Children's Oncology Group. Amifostine does not protect against the ototoxicity of high-dose cisplatin combined with etoposide and bleomycin in pediatric germ-cell tumors: a Children's Oncology Group study. Cancer. 2005 Aug 15;104(4):841-7. doi: 10.1002/cncr.21218. PMID 15999362